CLINICAL TRIAL: NCT02098226
Title: Method Comparison Protocol: MALDI Biotyper-Clinical Applications (MBT-CA) Phase 2
Brief Title: Evaluation of MALDI Biotyper CA System for Detection of Gram- and Gram+ Bacteria and Yeasts
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bruker Daltonics (Industry)
Responsible Party: Sponsor
Other Study IDs: BDAL-2013-001
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study objective is to confirm that the MBT-CA System identifies medically significant bacteria and yeasts from an isolated colony from any sample type processed by the clinical laboratory. For this purpose MBT-CA test results will be compared to bi-directional sequencing results.

DETAILED DESCRIPTION:
Bacteria or yeast isolates (1) fresh from primary culture plates, (2) collected directly from clinical samples, stored in the refrigerator or frozen or (3) well characterized organisms from a variety of contemporary culture collections will be included in the study. All organisms to be included in the study will be cultured on an agar medium prior to measurement.

Testing will be performed for various Gram negative and Gram positive bacteria and yeasts as outlined below. Several thousands of samples will be measured via MBT-CA systems based on MALDI-TOF MS technology (matrix assisted laser desorption ionisation time-of-flight mass spectrometry) at the test sites as fresh or frozen isolates of bacteria and yeasts. Lower prevalence organisms may be supplemented from banked culture collections.

The MBT-CA system uses an organism identification based on unique protein patterns of the microorganisms obtained from mass spectrometry. The test organism's spectrum (a pattern of mass peaks) is compared with a reference spectra library (database). Using biostatistical analysis, a probability ranking of the organism identification is generated. The probability ranking is represented as a log(score) between 0.00 and 3.00. Organism identification is reported with high confidence if the log(score) is ≥ 2.00. An organism identification is reported with low confidence if the log(score) is between 1.70 and <2.00.

In the last step the samples are sent to a special site for sequencing. Finally, the respective sequencing results are compared with the MBT-CA results.

Target microorganisms of study:

1. Acinetobacter haemolyticus
2. Acinetobacter johnsonii
3. Acinetobacter junii
4. Actinomyces meyeri
5. Actinomyces neuii
6. Actinomyces odontolyticus
7. Actinomyces oris
8. Aerococcus urinae
9. Aerococcus viridans
10. Aeromonas salmonicida
11. Anaerococcus vaginalis
12. Bacteroides fragilis
13. Bacteroides uniformis
14. Bacteroides_ovatus group
15. Bacteroides_thetaiotaomicron group
16. Bacteroides_vulgatus group
17. Bordetella group[3]
18. Bordetella hinzii
19. Brevibacterium casei
20. Brevundimonas_diminuta group
21. Campylobacter coli
22. Campylobacter jejuni
23. Campylobacter ureolyticus
24. Candida albicans
25. Candida boidinii
26. Candida dubliniensis
27. Candida duobushaemulonii
28. Candida famata
29. Candida glabrata
30. Candida guilliermondii
31. Candida haemulonis
32. Candida inconspicua
33. Candida kefyr
34. Candida krusei
35. Candida lambica
36. Candida lipolytica
37. Candida lusitaniae
38. Candida metapsilosis
39. Candida norvegensis
40. Candida orthopsilosis
41. Candida parapsilosis
42. Candida pararugosa
43. Candida pelliculosa
44. Candida tropicalis
45. Candida valida
46. Capnocytophaga ochracea
47. Capnocytophaga sputigena
48. Chryseobacterium gleum
49. Chryseobacterium indologenes
50. Clostridium difficile
51. Clostridium perfringens
52. Corynebacterium amycolatum
53. Corynebacterium bovis
54. Corynebacterium diphtheriae
55. Corynebacterium glucuronolyticum
56. Corynebacterium jeikeium
57. Corynebacterium kroppenstedtii
58. Corynebacterium macginleyi
59. Corynebacterium minutissimum
60. Corynebacterium propinquum
61. Corynebacterium pseudodiphtheriticum
62. Corynebacterium riegelii
63. Corynebacterium tuberculostearicum
64. Corynebacterium ulcerans
65. Corynebacterium urealyticum
66. Corynebacterium xerosis
67. Corynebacterium_aurimucosum group
68. Corynebacterium_striatum group
69. Cronobacter_sakazakii group
70. Cryptococcus gattii
71. Cryptococcus neoformans_var_grubii
72. Cryptococcus neoformans_var_neoformans
73. Cupriavidus_pauculus group
74. Delftia_acidovorans group
75. Dermacoccus nishinomiyaensis
76. Edwardsiella tarda
77. Elizabethkingia_meningoseptica group
78. Enterobacter amnigenus
79. Enterococcus casseliflavus
80. Enterococcus faecalis
81. Enterococcus faecium
82. Enterococcus gallinarum
83. Enterococcus hirae
84. Enterococcus_avium group
85. Finegoldia magna
86. Fusobacterium canifelinum
87. Fusobacterium necrophorum
88. Fusobacterium nucleatum
89. Gardnerella vaginalis
90. Gemella haemolysans
91. Gemella sanguinis
92. Geotrichum candidum
93. Geotrichum capitatum
94. Granulicatella adiacens
95. Haemophilus haemolyticus
96. Haemophilus influenzae
97. Haemophilus_parahaemolyticus group
98. Kingella kingae
99. Kloeckera apiculata
100. Kocuria kristinae
101. Kytococcus sedentarius
102. Lactococcus garvieae
103. Lactococcus lactis
104. Leuconostoc mesenteroides
105. Macrococcus caseolyticus
106. Micrococcus luteus
107. Moraxella_sg_Moraxella nonliquefaciens
108. Myroides odoratimimus
109. Myroides odoratus
110. Oligella ureolytica
111. Oligella urethralis
112. Parabacteroides distasonis
113. Pediococcus pentosaceus
114. Peptoniphilus_harei group
115. Peptostreptococcus anaerobius
116. Pichia ohmeri
117. Plesiomonas shigelloides
118. Porphyromonas gingivalis
119. Prevotella bivia
120. Prevotella buccae
121. Prevotella denticola
122. Prevotella intermedia
123. Prevotella melaninogenica
124. Propionibacterium acnes
125. Pseudomonas stutzeri
126. Rhizobium radiobacter
127. Rothia aeria
128. Rothia dentocariosa
129. Rothia mucilaginosa
130. Saccharomyces cerevisiae
131. Serratia plymuthica
132. Serratia rubidaea
133. Staphylococcus aureus
134. Staphylococcus auricularis
135. Staphylococcus capitis
136. Staphylococcus caprae
137. Staphylococcus carnosus
138. Staphylococcus cohnii
139. Staphylococcus epidermidis
140. Staphylococcus equorum
141. Staphylococcus felis
142. Staphylococcus haemolyticus
143. Staphylococcus hominis
144. Staphylococcus lugdunensis
145. Staphylococcus pasteuri
146. Staphylococcus pettenkoferi
147. Staphylococcus pseudintermedius
148. Staphylococcus saccharolyticus
149. Staphylococcus saprophyticus
150. Staphylococcus schleiferi
151. Staphylococcus simulans
152. Staphylococcus vitulinus
153. Staphylococcus warneri
154. Streptococcus agalactiae
155. Streptococcus anginosus
156. Streptococcus constellatus
157. Streptococcus dysgalactiae
158. Streptococcus gallolyticus
159. Streptococcus gordonii
160. Streptococcus intermedius
161. Streptococcus lutetiensis
162. Streptococcus mutans
163. Streptococcus pneumoniae
164. Streptococcus pyogenes
165. Streptococcus salivarius
166. Streptococcus_mitis_oralis group
167. Sutterella wadsworthensis
168. Trichosporon asahii
169. Vibrio parahaemolyticus
170. Vibrio vulnificus

sg = subgenus sp=species var = variety

ELIGIBILITY:
Inclusion Criteria:

-Patients with infections from certain yeasts, Gram positive or Gram negative bacteria (see Detailed Description)

Exclusion Criteria:

-Patients without infections from the quoted microorganisms (see Detailed Description)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with infections from certain yeasts, Gram positive or certain Gram negative bacteria (see Further Information / Target microorganisms of study)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Substantial equivalence of MBT-CA with sequencing concerning determination of the respective bacteria and yeasts | half a year

CONTACTS AND LOCATIONS:
Locations (1):
- Bruker Daltonik GmbH, Bremen, City state Bremen, Germany